CLINICAL TRIAL: NCT02183961
Title: Comparison of Three Methods Used in the Diagnosis of Extraesophageal Reflux in Children With Chronic Otitis Media With Effusion
Brief Title: Three Methods Used in the Diagnosis of EER in Children With OME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-EER Peptest Restech
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Otitis Media With Effusion; Laryngopharyngeal Reflux
Keywords: otitis media with effusion; peptest; restech; oropharyngeal pH monitoring; laryngopharyngeal reflux
MeSH Terms: conditions — Otitis Media with Effusion; Laryngopharyngeal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laryngopharyngeal reflux (Experimental): EER was detected using three methods: oropharyngeal pH was monitored for 24 hours using the Restech system; detection of pepsin in middle ear fluid obtained during myringotomy was done using Peptest, and detection of pepsin in adenoid specimen was done immunohistochemically using antibody P3635Rb-h.
  Interventions: Other: Restech; Other: Peptest; Other: Detection of pepsin in adenoid specimen

INTERVENTIONS:
Other: Restech
Other: Peptest
Other: Detection of pepsin in adenoid specimen

SUMMARY:
Detection of extraesophageal reflux (EER) in children with chronic otitis media with effusion (OME) using three different diagnostic methods and selection of the group of patients with severe EER who could potentially benefit from antireflux therapy.

DETAILED DESCRIPTION:
Children aged between 1 and 7 years diagnosed with bilateral or unilateral OME who underwent adenoidectomy and myringotomy with insertion of a ventilation tube were included in the prospective study. OME was defined as effusion in the middle ear behind an intact eardrum for longer than 3 months. Diagnosis was made on the basis of otomicroscopic findings, pneumatic otoscopy, type B tympanometry and audiometry (in older, cooperative children). Children with no fluid in the middle ear during myringotomy were re-diagnosed as having tympanosclerosis and were excluded from the study. Children with craniofacial abnormalities (Down syndrome, Treacher Collins syndrome, clefts etc.) were excluded from the study as well. Demographic data and symptoms of EER disease were provided by parents, who were specifically asked about hoarseness, recurrent lower respiratory infections (bronchitis, pneumonia) and bronchial asthma in their child.

24 hour monitoring of oropharyngeal pH using the Restech system was performed before surgery. Parents were instructed to record the time their child spent eating, drinking and in a horizontal position directly to the device and manually to the diary. If there was any discrepancy, periods logged in the device were modified according to the diary. A standardized RYAN composite score was calculated automatically using the software supplied. Patients with pathological RYAN composite scores in the vertical (higher than 9.4) and/or horizontal (higher than 6.8) position were classified as having pathological EER. Severe EER was diagnosed when the RYAN composite score in the vertical or horizontal position was higher than 200.

Myringotomy using a microscope was done on the anterior inferior part of the tympanic membrane. The type of middle ear effusion (fluid, mucous) was registered. Middle ear fluid was collected using a special suction device with a collecting bottle, and a ventilation tube was inserted in the tympanic membrane. In the case of bilateral OME, middle ear fluids were collected and analysed separately. The specimen was first standardized. 0.1 ml of 10% citric acid was added, the specimen was centrifuged for 10 minutes and subsequently the original migration reagent was added. Afterwards, the specimen was examined using Peptest, which contains monoclonal antibodies that target pepsin. The result of the Peptest was given as positive (2 lines), negative (1 line) or invalid (no line).

Then, adenoidectomy using a cold instrument was performed. A specimen of adenoids (5x5x5mm) from the area close to the torus tubarius was fixed in formaldehyde and immunohistochemically analysed at the Department of Pathology. Antibody P3635Rb-h (Uscnlife, USA, concentration 1:100) was used as the primary antibody. Antibody N-HistofineSimple Stain MAX PO (Nichirei Biosciences Inc.) was used as the secondary antibody.

Statistical analysis was done using MS Excel.

ELIGIBILITY:
Inclusion Criteria:

* children with otitis media with effusion
* age 1-7 years
* signing of the informed consent

Exclusion Criteria:

- children with craniofacial abnormalities (Down syndrome, Treacher Collins syndrome, clefts etc.)

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The frequency of the extraesophageal reflux in children with otitis media with effusion measured with three different methods | 2 years
  Children between 1 to 7 years diagnosed with OME who underwent adenoidectomy and myringotomy with insertion of a ventilation tube were included in this prospective study. EER was detected using three methods: oropharyngeal pH was monitored for 24 hours using the Restech system; detection of pepsin in middle ear fluid obtained during myringotomy was done using Peptest, and detection of pepsin in an adenoid specimen was done immunohistochemically using antibody P3635Rb-h.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Formánek, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] O'Reilly RC, He Z, Bloedon E, Papsin B, Lundy L, Bolling L, Soundar S, Cook S, Reilly JS, Schmidt R, Deutsch ES, Barth P, Mehta DI. The role of extraesophageal reflux in otitis media in infants and children. Laryngoscope. 2008 Jul;118(7 Part 2 Suppl 116):1-9. doi: 10.1097/MLG.0b013e31817924a3. PMID 18594333
- [Background] Zelenik K, Matousek P, Urban O, Schwarz P, Starek I, Kominek P. Globus pharyngeus and extraesophageal reflux: simultaneous pH <4.0 and pH <5.0 analysis. Laryngoscope. 2010 Nov;120(11):2160-4. doi: 10.1002/lary.21147. PMID 20938965
- [Background] Jiang A, Liang M, Su Z, Chai L, Lei W, Wang Z, Wang A, Wen W, Chen M. Immunohistochemical detection of pepsin in laryngeal mucosa for diagnosing laryngopharyngeal reflux. Laryngoscope. 2011 Jul;121(7):1426-30. doi: 10.1002/lary.21809. Epub 2011 Jun 6. PMID 21647907
- [Background] Wiener GJ, Tsukashima R, Kelly C, Wolf E, Schmeltzer M, Bankert C, Fisk L, Vaezi M. Oropharyngeal pH monitoring for the detection of liquid and aerosolized supraesophageal gastric reflux. J Voice. 2009 Jul;23(4):498-504. doi: 10.1016/j.jvoice.2007.12.005. Epub 2008 May 12. PMID 18468849